CLINICAL TRIAL: NCT02114476
Title: Effect of Implantable Progestin-only Contraception on the Incidence of Type 2 Diabetes and Metabolic Syndrome in Thai Women With History of Gestational Diabetes
Brief Title: Effect of Implantable Contraception on Type-2 DM and Metabolic Syndrome in Women With History of Gestational DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Manee Rattanachaiyanont, Department of Obstetrics and Gynecology, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GDM-Imp
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus; Metabolic Syndrome
Keywords: GDM; implant; diabetes mellitus; metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nonhormonal contraception (Placebo Comparator): nonhormonal intrauterine device tubal sterilization
  Interventions: Device: Placebo
- progestin implant (Experimental): Jadelle
  Interventions: Device: progestin implant

INTERVENTIONS:
Device: progestin implant — two small (2.5 mm × 43 mm) silicone rods each containing 75 mg of levonorgestrel in a polymer matrix
  Other Names: Jadelle
  Arms: progestin implant
Device: Placebo
  Arms: nonhormonal contraception

SUMMARY:
The purpose of this study is to determine the effect of implantable contraception on the incidence of diabetes mellitus in women with history of gestational diabetes mellitus comparing with those using nonhormonal contraceptives.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) was defined as abnormal glucose tolerance detected for the first time in pregnancy. GDM is a well-known risk factor for developing overt diabetes later in life, especially type 2 diabetes. About 50-60% of woman with prior GDM will develop type 2 diabetes during their lifetime. Recent studies show that women with previous GDM exhibit a markedly increased prevalence of the metabolic syndrome, even when glucose tolerance is normal. For both maternal and future offspring, women with prior GDM need safe, efficient, and acceptable choices for contraceptive methods that do not enhance their already substantial risk to develop either overt diabetes or metabolic syndrome and associated sequelae. The intrauterine device (IUD) is a very effective and reversible contraceptive method without metabolic disturbances and therefore is an ideal contraceptive for women with prior GDM. Progestins do not increase globulin production; thus, they do not increase coagulation factors or blood pressure. A nonrandomized open-label prospective trial of healthy obese, reproductive-age women in California were studied about the metabolic effects of progestin-only long-acting reversible contraception levonorgestrel-releasing intrauterine system (LNG-IUS) and etonogestrel implant (ENG-I)] comparing with nonhormonal contraception (NHC). The changes in fasting glucose and insulin sensitivity were seen among obese at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women with diagnosis of gestational diabetes mellitus
* Want to use implant contraception or nonhormonal contraceptions such as IUD or tubal sterilization

Exclusion Criteria:

* Age less than 18 years old
* Diagnosis of diabetes mellitus at post partum period
* Cardiovascular disease, Liver disease, autoimmune disease
* The women that reject to continue in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Diabetes mellitus | 5 years
  Incidence of type-2 DM in women with history of gestational diabetes using implantable contraception.

SECONDARY OUTCOMES:
metabolic syndrome | 5 years
  Prevalence of metabolic syndrome in women with history of gestational diabetes using implantable contraception.

CONTACTS AND LOCATIONS:
Overall Officials: Manee Rattanachaiyanont, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand